CLINICAL TRIAL: NCT07134543
Title: Using the Smart Underwear Device to Determine a Baseline of Flatus Activity Normalized to Fiber Intake
Status: Recruiting | Type: Observational
Sponsor: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Other Study IDs: Human Flatus Atlas
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: All Health Backgrounds to Determine a Baseline of Flatus Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- American adults: American adults that are at least 18 years old, live in the United States, are not pregnant or lactating, and agree to wear the Smart Underwear device.

SUMMARY:
The goal of this observational study is to quantify the typical frequency of flatulence in healthy adults, normalized by fiber intake, using the Smart Underwear device. The study will enroll a maximum of 500 adults across the United States who will wear the device for three consecutive days while continuing their usual daily activities.

The main questions it aims to answer are:

* What is the average frequency of flatus events in a general adult population?
* How does dietary fiber intake influence flatus frequency and microbiome activity?

Researchers will collect gas sensor data from the Smart Underwear device alongside dietary information logged in a mobile app to assess the relationship between diet and microbiome activity.

Participants will:

* Complete an online eligibility survey, consent form, and background questionnaire.
* Wear the Smart Underwear device for at least 12 hours per day for three consecutive days.
* Log all meals with photos using a custom smartphone app.
* Complete a short post-wear survey about device comfort and usability.

All study procedures will be conducted remotely. Data will be analyzed in de-identified form to evaluate baseline flatulence patterns, normalized to fiber intake, in the general adult population.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Lives in the US
* Is not pregnant or lactating
* Is willing to wear the Smart Underwear device as instructed in the study procedures

Exclusion Criteria:

* Younger than 18 years old
* Lives outside the US
* Is pregnant or lactating
* Is not willing to wear the Smart Underwear device as instructed in the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of the US
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-09-05 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Microbiome Activity Index | 12 hours each day for 3 days
  The Microbiome Activity Index is a composite measure reflecting gut microbiome activity, calculated from both flatus frequency and hydrogen gas concentration. The index uses the absolute value of the first derivative of the hydrogen sensor signal to better capture flatus intensity, reduce baseline noise, and mitigate sensor saturation at high hydrogen levels. This composite approach ensures a more accurate representation of gut microbiome activity than relying on flatus count or hydrogen concentration alone. Data are collected using a wearable device ("Smart Underwear") and uploaded to the Human Flatus Atlas app.

SECONDARY OUTCOMES:
Total flatus count | 12 hours each day for 3 days
  The total number of flatus events detected by the wearable device. Detection is based on hydrogen gas concentration changes and signal rate-of-change analysis.
Flatus Per Hour | 12 hours each day for 3 days
  The rate of flatus events normalized per hour, calculated from the total number of events and the total monitored time.
Microbiome Activity Index Comparative Score | 12 hours each day for 3 days
  A relative score comparing the participant's Microbiome Activity Index to aggregated anonymized results from other individuals in the Human Flatus Atlas study. Presented as a percentile rank or standardized score.
Fiber-Normalized Flatus Frequency | 12 hours each day for 3 days
  The participant's flatus frequency (events/day) normalized by self-reported dietary fiber intake (grams/day). Normalization will allow assessment of typical adult flatulence frequency in relation to fiber consumption.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Bioscience Research Building, College Park, Maryland
  - University of Maryland Bioscience Research Building, College Park, Maryland

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified, aggregate individual participant data limited to total enrollment numbers and demographic characteristics (e.g., age range, sex distribution, and other baseline variables) collected during the study. No other data, including outcome or clinical data, will be shared.
  Supporting Information The shared dataset will not contain any information that could directly or indirectly identify participants. Data will be available in aggregate format only, and will be provided upon reasonable request from qualified researchers for the purposes of scientific transparency and verification of study population characteristics.
Supporting Information: Study Protocol